CLINICAL TRIAL: NCT05402293
Title: Pharmacokinetic Profile of Lidocaine Given as a Weight-based Infusion for Postoperative Surgical Pain Control
Status: Terminated | Type: Observational
Why Stopped: Enrollment difficulties
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00089761
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Pain; Lidocaine; Administration and Dosage
Keywords: Acute Pain; Lidocaine Infusion; Pharmakokinetics; Post-operative analgesia
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — Plasma samples for analysis of lidocaine concentration Will be disposed of following analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Blood samples to measure lidocaine levels — Blood sampling is the only intervention Plasma samples will then be analyzed for lidocaine concentration

SUMMARY:
Study Summary

Title Pharmacokinetic profile of lidocaine given as a weight-based infusion for postoperative surgical pain control

Short Title Pharmacokinetic profile of lidocaine given as a weight-based infusion for postoperative surgical pain control

Methodology Pharmacokinetic study of lidocaine in the surgical population

Study Duration 1 year

Study Center(s) University of Alberta Hospital

Objectives The primary objective will be to map serum lidocaine levels over time in a diverse surgical patient population receiving a weight-based lidocaine infusion.

Number of Subjects 40

Diagnosis and Main Inclusion Criteria ASA class 1-3 Age 18-40 or >75 Scheduled for elective major ENT flap, urology or general surgery.

Study Product, Dose, Route, Regimen Lidocaine IV infusion

* 1.5mg/kg bolus, then
* 1mg/kg/h IV intraoperatively, then
* 0.5-2 mg/kg/hr IV for 48 h, depending on clinical response

DETAILED DESCRIPTION:
1. Background Information

1.1 Investigational Product Lidocaine HCl 2%, perioperative intravenous weight-based infusion over 48 h

1.2 Summary of Literature Given the ongoing opiate epidemic there is a need for alternative multimodal analgesia approaches to post-surgical pain. Intravenous lidocaine infusions are known to be effective for the management of acute perioperative pain,(1-5) and may help prevent the development of chronic pain(6). Guidelines have been developed to guide clinical practice (6) and lidocaine infusions are used routinely in many centres throughout Canada for post-surgical pain management.

The currently accepted plasma lidocaine levels required for acute analgesia are 1.1 - 4.2 μg/mL (7-9) with a tighter goal of 2.5 - 3.5 μg/mL recommended in other papers (6). Minor adverse CNS effects have been described at a plasma level of 5-10 μg/mL, with more serious CNS and CVS effects reported at levels greater than 10 μg/mL(6,7,9). Minor CNS effects therefore occur at levels outside but close to the upper limits of the described therapeutic ranges.

Current pharmacokinetic data used to guide lidocaine infusions have been derived largely from studies using healthy volunteers. Factors such as age, BMI and the stress response to surgery can alter pharmacokinetics via mechanisms including altered hepatic blood flow and changes in serum proteins(6-8,12). Accurate pharmacokinetic modelling of weight-based lidocaine infusions in elderly patients and in those with higher BMI following major surgery is incomplete however and detailed pharmacokinetic data for these patient groups is required to optimize safe and effective analgesia.

The study proposes to collect data to accurately model lidocaine pharmacokinetics in the post-surgical population. We hypothesise that weight-based pharmacokinetics will yield a predictable lidocaine concentration with possible outliers being morbidly obese patients and the elderly.

1.3 Risk/Benefits Multimodal analgesia is standard of care for patients undergoing major surgery. Lidocaine infusion is one element of multimodal analgesia and can be used for patients undergoing major surgery both intra-operatively and postoperatively. Options for multimodal analgesia are discussed with patients pre-operatively in the pre-operative anesthetic assessment clinic and on the day of surgery with the anesthetist and the Acute Pain Service team. Only patients suitable for lidocaine infusion who have agreed to this as part of their multimodal analgesia care will be eligible to be approached for study recruitment.

The study does not alter the type of analgesia drugs given as we will simply be collecting blood samples from patients already agreeing to have multimodal analgesia which includes lidocaine infusion. There is therefore no benefit to the patient to be enrolled in the study. The risks of study participation are discomfort and bruising from blood collection although we will try and reduce this by collecting blood samples through an existing IV cannula or arterial line.

1.4 Route, Dosage, Treatment Regimen Lidocaine infusions are given in line with the Ottawa protocol(6) including standard monitoring. Lidocaine will be given as a 1.5 mg/kg bolus (max 100mg) over 4 minutes, followed immediately by an infusion of 1 mg/kg/h intraoperatively and then titrated between 0.5-2 mg/kg/h for 48 h, by the Acute Pain Service depending on clinical response according to usual practice.

Venous blood samples (5 mL) will be drawn via the in-situ IV cannula or arterial line if one has been sited at 4 pre-set times, as well as immediately prior to any adjustment to the infusion level, and 4 hours after adjustment to the infusion levels.

1.5 Statement of Compliance This study will be conducted in compliance with the protocol approved by the University of Alberta Health Research Ethics Board (HREB), and according to Good Clinical Practice standards. No deviation from the protocol will be implemented without the prior review and approval of the HREB except where it may be necessary to eliminate an immediate hazard to a research subject. In such case, the deviation will be reported to the HREB as soon as possible. Contracts will be negotiated with NACTRC, and the trial will be registered with ClinicalTrials.gov.

1.6 Population

Inclusion criteria are:

* Age 18-40 or >75
* ASA 1-3
* Scheduled for elective major surgery at the University of Alberta Hospital in which lidocaine infusion would be a good option as part of standard multimodal analgesia care

Exclusion criteria:

* Contraindication / History of hypersensitivity to lidocaine or amide local anesthetics
* Inability to give informed consent (illiteracy, <7th grade education)
* NYHA class III-IV heart disease
* Planned epidural or regional anesthesia technique requiring local anesthetic

All patients filling the stated inclusion and exclusion criteria will be eligible and will be identified and approached for consent via the Pre-Admission Clinic prior to the day of surgery.

1.7 References

1. Khan JS, Yousuf M, Victor JC, Sharma A, Siddiqui N. An estimation for an appropriate end time for an intraoperative intravenous lidocaine infusion in bowel surgery: a comparative meta-analysis. J Clin Anesth. 2016 Feb;28:95-104.
2. Kim K-T, Cho D-C, Sung J-K, Kim Y-B, Kang H, Song K-S, et al. Intraoperative systemic infusion of lidocaine reduces postoperative pain after lumbar surgery: a double-blinded, randomized, placebo-controlled clinical trial. Spine J. 2014 Aug;14(8):1559-66.
3. Kranke P, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, et al. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery. Cochrane Anaesthesia, Critical and Emergency Care Group, editor. Cochrane Database Syst Rev [Internet]. 2015 Jul 16 [cited 2018 Oct 9]; Available from: http://doi.wiley.com/10.1002/14651858.CD009642.pub2
4. Weibel S, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, et al. Efficacy and safety of intravenous lidocaine for postoperative analgesia and recovery after surgery: a systematic review with trial sequential analysis † †This review is an abridged version of a Cochrane Review previously published in the Cochrane Database of Systematic Reviews 2015, Issue 7, DOI: CD009642 (see www.thecochranelibrary.com for information).1 Cochrane Reviews are regularly updated as new evidence emerges and in response to feedback, and Cochrane Database of Systematic Reviews should be consulted for the most recent version of the review. Br J Anaesth. 2016 Jun;116(6):770-83.
5. De Oliveira GS, Duncan K, Fitzgerald P, Nader A, Gould RW, McCarthy RJ. Systemic Lidocaine to Improve Quality of Recovery after Laparoscopic Bariatric Surgery: A Randomized Double-Blinded Placebo-Controlled Trial. Obes Surg. 2014 Feb;24(2):212-8.
6. Eipe N, Gupta S, Penning J. Intravenous lidocaine for acute pain: an evidence-based clinical update. BJA Educ. 2016 Sep;16(9):292-8.
7. Weinberg L, Peake B, Tan C, Nikfarjam M. Pharmacokinetics and pharmacodynamics of lignocaine: A review. World J Anesthesiol. 2015 Jul 27;4(2):17-29.
8. Hsu Y-W, Somma J, Newman M, Mathew JP. Population Pharmacokinetics of Lidocaine Administered During and After Cardiac Surgery. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):931-6.
9. Dewinter GBE, Teunkens A, Vermeulen K, Al tmimi L, Van de Velde M, Rex S. Systemic Lidocaine Fails to Improve Postoperative Pain, But Reduces Time to Discharge Readiness in Patients Undergoing Laparoscopic Sterilization in Day-Case Surgery: A Double-Blind, Randomized, Placebo-Controlled Trial. Reg Anesth Pain Med. 2016;41(3):362-7.
10. Yousefshahi F, Predescu O, Francisco Asenjo J. The Efficacy of Systemic Lidocaine in the Management of Chronic Pain: A Literature Review. Anesthesiol Pain Med [Internet]. 2017 Apr 22 [cited 2018 Oct 9];7(3). Available from: http://anesthpain.neoscriber.org/en/articles/55837.html
11. Cox B, Durieux ME, Marcus MAE. Toxicity of local anaesthetics. Best Pract Res Clin Anaesthesiol. 2003 Mar 1;17(1):111-36.
12. Daykin H. The efficacy and safety of intravenous lidocaine for analgesia in the older adult: a literature review. Br J Pain. 2017 Feb;11(1):23-31.
13. Al Nebaihi HM, Primrose M, Green JS, Brocks DR. A High-Performance Liquid Chromatography Assay Method for the Determination of Lidocaine in Human Serum. Pharmaceutics. 2017 Dec;9(4):52.

2 Trial Objectives and Purpose Lidocaine infusions are known to be effective for the management of acute perioperative pain and may help prevent the development of chronic pain. The currently accepted plasma lidocaine levels required for acute analgesia are between 1.1 - 4.2 mcg/mL. Minor adverse effects have been described at plasma levels as low as 5 mcg/mL which is just above the therapeutic range. Current pharmacokinetic data for lidocaine infusions have largely been derived from studies using healthy volunteers rather than in patients undergoing major surgery which can lead to error in predicting plasma levels. The primary objective of this cohort study is to accurately map serum lidocaine levels over time in patients undergoing major surgery. Age, sex and BMI will be used as covariates for sub analysis. This data will be valuable to increase the efficacy and safety of lidocaine infusions for the prevention and treatment of post-operative pain in patients undergoing major surgery.

3 Trial Design

3.1 Primary Study Endpoints/Secondary Endpoints Lidocaine infusions run as per Ottawa protocol for a maximum of 48 hours. Patient participation will end following the last blood draw which will take place 2-4 hours after discontinuation of lidocaine infusion.

Endpoints in this study will be pharmacological. The primary endpoint of this trial is the mapping of serum lidocaine levels over time in a diverse surgical patient population. Three covariates will be used for sub analysis: age, sex, and BMI. Data will be analysed in a group batch following collection of blood samples from all 40 study patients.

No secondary endpoints will be analysed in this study.

3.2 Study Design/Type Pharmacokinetic study of lidocaine in the surgical population. The study will include 40 patients, allocated by age, sex, and BMI in groups of 5.

Sex Age BMI Planned number of Patients

1 Male 18-40 <25 5 2 Male 18-40 >35 5 3 Female 18-40 <25 5 4 Female 18-40 >35 5 5 Male >75 <25 5 6 Male >75 >35 5 7 Female >75 <25 5 8 Female >75 >35 5

3.3 Randomization This trial is not randomized.

3.4 Trial Treatment Patients will receive standard CAS monitoring. Anesthetic choice will be left to the discretion of the attending anesthetist, with the exception of local anesthetic administration, which will be started according to the Ottawa standardized protocol intraoperatively: Induction will include a 1.5 mg/kg bolus of lidocaine (max 100mg) over 4 minutes intravenously, followed immediately by an infusion of 1 mg/kg/h intraoperatively and then titrated between 0.5-2 mg/kg/h for 48 h, by the Acute Pain Service depending on clinical response according to usual practice.

Venous blood samples (5 mL) will be drawn via the in-situ IV cannulae at 4 pre-set times, as well as immediately prior to any adjustment to the infusion level, and 4 hours after adjustment to the infusion levels. A population pharmacokinetic approach will be used to estimate the pharmacokinetic parameters of interest. This will require only sparse, rather than intensive, sampling of the patient's blood to obtain the pharmacokinetic data. Therefore, blood samples will be taken at the following pre-defined intervals:

* 10 - 30 min after bolus
* 2-6h after bolus
* Immediately before the end of the infusion
* 2-4 h after end of infusion
* Immediately prior to a change in the infusion level
* 4 h after a change in infusion level Samples will be immediately centrifuged and stored at -80C until analysis by liquid chromatography assay.

3.5 Duration Active subject participation is from the time of consent to 48 hours after surgery.

3.6 Discontinuation Each patient will receive standardized monitoring for Local Anesthetic Toxicity, as per hospital protocol. In the event of suspected Local Anesthetic Toxicity, the Acute Pain Services team and the study team will be advised, the lidocaine infusion will be discontinued immediately, and a venous sample will be drawn as per protocol. Additionally, each patient is free to withdraw from the trial at any time, after which no further data will be collected.

Beyond serum sample collection, medical treatment of subjects will be not be different from medical treatment if they were not included in the trial. As such, there are currently no criteria for termination of the trial beyond subject withdrawal.

3.7 Accountability procedures

Intravenous lidocaine is currently used in daily practice in our institution. Vials of 1% and 2% lidocaine are available for use in anesthetic drug carts positioned in the operating room theatres, and in the block area used by the acute pain service team. Pharmacy prepares 0.4% lidocaine in 250mls bags for low dose lidocaine infusions intended for use in post-operative pain management.

As such, use of the investigational product (Lidocaine) is not restricted to the study and no special provision for storage will be required.

Lidocaine use and protocol adherence will be verified by examination of the patient electronic medical records.

This study will not use placebo or comparators.

3.8 Data Identification Collection of the patient's name and health care number will be necessary to track patients through their operation and hospitalization. This information will be removed prior to entry in the clinical database.

All identifying information will be removed by the research coordinator prior to entry into a clinical database. Personal identifiers will be destroyed following the 48-hour serum sampling timeframe. A key will be kept by the research coordinator separately and this will be destroyed once the study analysis is complete.

4 Selection and Withdrawal of Subjects

4.1 Inclusion Criteria

* Age 18-40 or >75
* ASA 1-3
* Scheduled for elective major surgery at the University of Alberta Hospital

4.2 Exclusion Criteria

* Contraindication / History of hypersensitivity to lidocaine or amide local anesthetics
* Inability to give informed consent (illiteracy, <7th grade education)
* NYHA class III-IV heart disease
* Planned epidural or regional anesthesia technique requiring local anesthetic

4.3 Subject Withdrawal Subjects may withdraw from the study at any time prior to or after the surgery by voicing that desire to any of the study investigators, without impact to their care. No attempts will be made to collect additional follow-up data from participants who have withdrawn consent.

Attempts where possible will be made to replace any withdrawn subjects with a further suitable candidate matching to the same cohort.

5 Treatment of Subjects

5.1 Treatment to be administered Patients will receive standard CAS monitoring. Anesthetic choice will be left to the discretion of the attending anesthetist, with the exception of local anesthetic administration, which will be standardized to the study protocol. As such, the induction will include a 1.5 mg/kg bolus of lidocaine over 4 minutes intravenously, followed immediately by an infusion (pumped at a flow rate to deliver 1 mg/kg/h for intraoperatively and then 0.5-2 mg/kg/h for 48 h, depending on clinical response - adjusted by the acute pain service according to usual practice).

5.2 Medications permitted and not permitted Anesthetic choice will be left to the discretion of the attending anesthetist, with the exception of local anesthetic.

5.3 Compliance monitoring The medications will be administered and monitored by researchers and the acute pain service. As such, no further procedures to monitor subject compliance are required.

6 Assessment of Efficacy

6.1 Efficacy Parameters The primary measured parameter will be serum lidocaine levels over time. The primary pharmacokinetic measures derived from those parameters will be clearance and volume of distribution. Half-life will also be determined. The measure of exposure will be the maximum and the steady state serum concentrations.

6.2 Method and Timing Venous blood draws (5-10 mL) will be done by the attending anesthesiologist intra-operatively, and by study investigators post-operatively.

Blood draws will be from the in-situ IV canulae.

A population pharmacokinetic approach using nonlinear mixed effects modelling will be used to estimate the lidocaine pharmacokinetic parameters of interest (maximal concentration after dosing, area under the concentration vs. time curve, clearance, volume of distribution, terminal phase half-life). This will require only sparse, rather than intensive, sampling of the patient's blood to obtain the pharmacokinetic data. Therefore, blood will be taken at the following intervals:

- 10-30 min after bolus

* 2-6h after bolus
* Immediately before the end of the infusion
* 2-4h after the end of the infusion
* Immediately prior to a change in the infusion level
* 4 h after a change in infusion level.

Samples will be immediately centrifuged and stored at -80C until analysis by liquid chromatographic assay. Precise timing of dose administration and blood sampling will be performed (to the nearest minute). A validated chromatographic assay will be used to measure lidocaine concentrations in the blood fluid specimens.(13)

7 Assessment of Safety

7.1 Safety Parameters Markers of intervention safety will be monitored include local anesthetic toxicity, hypersensitivity reactions.

7.2 Method and Timing The principle investigator and resident investigator will review any patient with signs or symptoms of local anesthetic toxicity.

7.3 Adverse Event Reporting Adverse event reporting will be in compliance with the University of Alberta HREB and Health Canada requirements.

The principle investigator or resident investigator will report any events that:

* impact the rights, safety or well-being of a research participant. Examples may include: enrolment of subject that does not meet the inclusion/exclusion criteria of the protocol, consent violations, subject visits which occur prior to study approval, or after expiry of study approval;
* jeopardize the study efficacy or the data integrity. Examples include significant variance from the protocol required study procedures; OR
* constitute a breach of privacy. All Serious Unexpected Adverse Drug Reactions will be reported to Health Canada, in accordance with Adverse Drug Reactions (ADRs) Reporting Criteria and Protocols, as outlined in sections 2.8.4.1 - 2.8.4.3 in Health Canada's Guidance Document for Clinical Trial Sponsors: Clinical Trial Applications. As per requirements, all ADRs meeting the criteria of serious, unexpected and suspected causal relationship will be reported.

7.4 Follow-up after adverse events Each patient will receive standardized monitoring for Local Anesthetic Toxicity, as per hospital protocol. In the event of suspected Local Anesthetic Toxicity, the Acute Pain Services team and the study team will be advised, the lidocaine infusion will be discontinued immediately, and a venous sample will be drawn as per protocol.

8 Statistical Plan

8.1 Statistical Methods Population pharmacokinetics No interim analysis is planned.

8.2 Number of subjects 40

8.3 Level of significance N/A in pharmacokinetic study

8.4 Criteria for termination of trial This study uses a drug, route, and dosage already employed in common practise. Beyond serum sample collection, medical treatment of subjects will be not be different from medical treatment if they were not included in the trial. As such, there are no criteria for termination of the trial beyond subject withdrawal.

8.5 Procedure for accounting for missing, unused and spurious data All pharmacokinetic data will be analysed and reported

8.6 Procedure for reporting deviations from original statistical plan N/A: This is a pharmacological study and all results will be reported in full

8.7 Selection of included subjects All subjects deemed eligible, having consented to the study, and where lidocaine infusion was initiated will have blood samples drawn and all of these will be included in the analysis.

9 Direct Access to Source Data/Documentation The investigators will permit trial-related monitoring, audits, HREB review and regulatory inspection(s) by providing direct access to source data/documentation.

10 Quality Control and Quality Assurance The principle investigator will ensure that the study will be conducted in compliance with Good Clinical Practice.

11 Ethical Considerations This study will be conducted according to Canadian and international standards of Good Clinical Practice for all studies. Applicable government regulations and University of Alberta research policies and procedures will also be followed.

This protocol and any amendments will be submitted to the University of Alberta HREB for formal approval to conduct the study.

All subjects for this study will be provided a consent form describing this study and providing sufficient information for subjects to make an informed decision about their participation in this study. This consent form will be submitted with the protocol for review and approval by the HREB. The formal consent of a subject, using the HREB-approved consent form, will be obtained before that subject is submitted to any study procedure. This consent form must be signed by the subject or legally acceptable surrogate, and the investigator-designated research professional obtaining the consent.

12 Data Handling and Record Keeping At no time will any patient information be distributed or left in public spaces. Patients will not be identified in any presentation or publication and no agencies or individuals outside of this research team will have access to the confidential data for this study now or in the future. All identifying information will be removed prior to the creation of the database and entered into a separate 'key' file. This key will be destroyed after completion of the study. Personal identifiers will be destroyed following the 48h serum sampling timeframe.

The principal investigator will communicate both prior to initiation of the trial, and throughout with members of the research team. Members of the research team that have access to data consist of physicians and nurses who have had training regarding privacy in their respective professions.

All records pertaining to this trial will be retained for a period of 25 years.

13 Finance and Insurance This study is not funded.

14 Publication Policy Will be submitted to a peer review journal.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1-3. Age 18-40 or >75. - Scheduled for elective major surgery at the University of Alberta Hospital in which lidocaine infusion would be a good option as part of standard multimodal analgesia care

Exclusion Criteria:

* Contraindication / History of hypersensitivity to lidocaine or amide local anesthetics
* Inability to give informed consent (illiteracy, <7th grade education)
* NYHA class III-IV heart disease
* Planned epidural or regional anesthesia technique requiring local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major elective surgery at the University of Alberta Hospital. Edmonton who are receiving lidocaine infusion as part of their post-operative pain management
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Lidocaine concentrations from plasma samples | 48 hours from initiation of lidocaine infusion
  The study will measure lidocaine concentrations in this surgical population receiving lidocaine infusion for post-operative analgesia

CONTACTS AND LOCATIONS:
Overall Officials: James Green, MB BS, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
The lidocaine concentration data will be presented in full in the published manuscript